CLINICAL TRIAL: NCT03122886
Title: Double-Blinded, Placebo-Controlled Pilot Trial to Explore Whether Lipids Prevent Carboplatin and Oxaliplatin Hypersensitivity Reactions
Brief Title: Fat Emulsion in Preventing Hypersensitivity Reactions in Patients With Cancer Receiving Carboplatin or Oxaliplatin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MC16C1; NCI-2017-00495 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC16C1 (Other: Mayo Clinic); UG1CA189823 (NIH); 16-007773 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2017-03-28; First posted 2017-04-21 (Actual); Results first posted 2020-05-20 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Advanced Malignant Neoplasm
MeSH Terms: interventions — soybean oil, phospholipid emulsion; Fat Emulsions, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (fat emulsion) (Experimental): Patients receive fat emulsion IV immediately before each dose of either carboplatin or oxaliplatin. Treatment continues for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: Fat Emulsion
- Group II (placebo) (Placebo Comparator): Patients receive placebo IV immediately before each dose of either carboplatin or oxaliplatin. Treatment continues for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Fat Emulsion — Given IV
  Other Names: FAT EMULSION, INTRAVENOUS; Intralipid; Intravenous Fat Emulsion
  Arms: Group I (fat emulsion)
Other: Placebo — Given IV
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Group II (placebo)

SUMMARY:
This randomized pilot trial studies how well fat emulsion works in preventing hypersensitivity reactions in patients with cancer receiving carboplatin or oxaliplatin. Giving lipids before chemotherapy may prevent some drug reactions from carboplatin or oxaliplatin.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the infusion of a lipid emulsion before each dose of chemotherapy appears to prevent carboplatin and oxaliplatin hypersensitivity reactions in high-risk patients.

II. To explore if lipid infusions modulate a well-established panel of mediators of hypersensitivity reactions and if these mediators appear to predict reactions.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive fat emulsion intravenously (IV) immediately before each dose of either carboplatin or oxaliplatin. Treatment continues for up to 2 years in the absence of disease progression or unacceptable toxicity.

GROUP II: Patients receive placebo IV immediately before each dose of either carboplatin or oxaliplatin. Treatment continues for up to 2 years in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Advanced, incurable cancer
* 7th or later cycle of intravenous carboplatin or oxaliplatin infusion planned or 4 months after the first cycle of agent (whichever is of longer duration) =< 30 days after registration
* Anticipated 2 or more subsequent chemotherapy infusions of either carboplatin or oxaliplatin at the time of study registration; NOTE: the dose of carboplatin or oxaliplatin, choice of other chemotherapy, and other ancillary treatment, such as antiemetics, will be left to the discretion of the treating healthcare provider
* Willing to provide mandatory blood and urine specimens for correlative research; NOTE: can be waived with permission of study chair (documentation such as an email must be provided)
* Serum creatinine =< 1.5 times the institutional upper limit of normal (ULN); NOTE: can be waived with permission of study chair (documentation such as an email must be provided)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 3 x the upper limit of normal
* Triglycerides < 500 mg/dL
* Alkaline phosphatase =< 3 x the institutional upper limit of normal

Exclusion Criteria:

* Concurrent liposomal doxorubicin or any other liposomal agent
* Prior carboplatin or oxaliplatin hypersensitivity reaction
* Taking aspirin, nonsteroidal anti-inflammatory agents, or zileuton =< 7 days prior to registration; NOTE: can be waived with permission of study chair (documentation such as an email must be provided)
* Allergy to egg or egg byproducts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group I (Fat Emulsion) | Group II (Placebo)
Started | 10 | 9
Completed | 9 | 7
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (Fat Emulsion) | Group II (Placebo) | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Median (Full Range); unit: years] | 67.5 [45 to 76] | 66 [44 to 80] | 66 [44 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 8 | 3 | 11
    1 | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Time-to-carboplatin or Oxaliplatin Acute Hypersensitivity Reaction
Description: The primary endpoint is the time to healthcare provider reported hypersensitivity reactions from either carboplatin or oxaliplatin. Kaplan Meier curves will be constructed and a log-rank test will be used to compare time-to-hypersensitivity reaction between treatment arms. Data will be censored based on last infusion with no hypersensitivity reaction with a maximum study treatment duration of 2 years per patient.
Time Frame: Up to 2 years
Population: Evaluable participants are included in this analysis (i.e. exclude Withdrawals).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group I (Fat Emulsion) | Group II (Placebo)
Number analyzed (Participants) | 9 | 7
months | 4.4 [1.4 to 4.4] | NA [2.8 to NA] — The median and 95% confidence interval upper limit was not evaluable (i.e. insufficient number of events observed to ascertain these summary statistics).
Statistical Analysis 1: Comparison: Group I (Fat Emulsion) vs Group II (Placebo); Test type: Superiority; p = 0.90, Log Rank; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.12 to 6.37]

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Evaluable participants are included in this analysis (i.e. exclude Withdrawals).
Arm/Group | Group I (Fat Emulsion) | Group II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/9 | 2/7
Other Adverse Events (participants affected / at risk) | 4/9 | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Fat Emulsion) (N=9) | Group II (Placebo) (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gen disord and admin site conds-Oth spec (General disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Fat Emulsion) (N=9) | Group II (Placebo) (N=7)
Allergic reaction (Immune system disorders) | 3 (3) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (4) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/86/NCT03122886/Prot_SAP_000.pdf